CLINICAL TRIAL: NCT00000745
Title: A Phase I Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of HIV-1 Recombinant Envelope Glycoprotein gp160
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 003; 10540 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Vaccines; HIV-1; HIV Envelope Protein gp160; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia | interventions — Hepatitis B Vaccines; VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: Hepatitis B Vaccine (Recombinant)
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
To determine the reactivity and safety of HIV-1 recombinant envelope glycoprotein gp160. To determine the immunogenicity of gp160.

Although recent advances have been made in antiviral therapy against AIDS, there is currently no cure. It is likely that ultimate control of the disease will depend on the development of safe and effective vaccines against HIV.

DETAILED DESCRIPTION:
Although recent advances have been made in antiviral therapy against AIDS, there is currently no cure. It is likely that ultimate control of the disease will depend on the development of safe and effective vaccines against HIV.

Healthy volunteers are injected on days 0, 30, and 180 with one of four preparations: gp160 vaccine (40 mcg), gp160 vaccine (80 mcg), hepatitis B vaccine, and placebo. The hepatitis B vaccine group will serve as an additional control for immunological evaluations. An optional fourth injection may be given 15-21 months following the initial inoculation.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* Negative for HIV infection by ELISA and Western blot (i.e., no reactivity at gp160, gp120, gp41, or p24).
* T4 count >= 800 cells/mm3.
* Normal chest x-ray and urinalysis.
* Negative surface antibody and core antibody for hepatitis B.
* Negative hepatitis B surface antigen.
* Negative HIV p24 antigen test.
* Normal skin reactivity by Merieux test.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Positive PPD.
* Syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease).

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, or use of immunosuppressive medications.
* Prior hepatitis B vaccination.
* Syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease) in the past 6 months.

Prior Medication:

Excluded:

* Prior hepatitis B vaccine.

Prior Treatment:

Excluded:

* Prior blood transfusions or cryoprecipitates within the past 6 months.

Identifiable high-risk behavior for HIV infection (as determined by prescreening questions designed to identify risk factors for HIV infection), including:

* Any history of IV drug use.
* Syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease) in the past 6 months.
* More than two sexual partners, or sexual contact with a high-risk partner, in the past 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72
Dates: Study Completion 1991-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belshe R, Study Chair; Clements ML, Study Chair; Couch R, Study Chair; Dolin R, Study Chair; Levine M, Study Chair; Wright P, Study Chair
Locations (2):
- United States (2):
  - JHU AVEG, Pittsburgh, Pennsylvania
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee

REFERENCES:
- [Background] Dolin R, Graham BS, Greenberg SB, Tacket CO, Belshe RB, Midthun K, Clements ML, Gorse GJ, Horgan BW, Atmar RL, et al. The safety and immunogenicity of a human immunodeficiency virus type 1 (HIV-1) recombinant gp160 candidate vaccine in humans. NIAID AIDS Vaccine Clinical Trials Network. Ann Intern Med. 1991 Jan 15;114(2):119-27. doi: 10.7326/0003-4819-114-2-119. PMID 1984386
- [Background] Archibald DW, Hebert CA, Sun D, Tacket CO. Salivary antibodies to human immunodeficiency virus type 1 in a phase I AIDS vaccine trial. J Acquir Immune Defic Syndr (1988). 1990;3(10):954-8. PMID 2204698
- [Background] Westblom TU, Belshe RB, Gorse GJ, Anderson EL, Berry CF. Characteristics of a population volunteering for human immunodeficiency virus immunization. NIAID AIDS Clinical Trials Network. Int J STD AIDS. 1990 Mar;1(2):126-8. doi: 10.1177/095646249000100211. PMID 2092787
- [Background] Keefer MC, Wolff M, Gorse GJ, Graham BS, Corey L, Clements-Mann ML, Verani-Ketter N, Erb S, Smith CM, Belshe RB, Wagner LJ, McElrath MJ, Schwartz DH, Fast P. Safety profile of phase I and II preventive HIV type 1 envelope vaccination: experience of the NIAID AIDS Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 1997 Sep 20;13(14):1163-77. doi: 10.1089/aid.1997.13.1163. PMID 9310283
- [Background] Tacket CO, Baqar S, Munoz C, Murphy JR. Lymphoproliferative responses to mitogens and HIV-1 envelope glycoprotein among volunteers vaccinated with recombinant gp160. AIDS Res Hum Retroviruses. 1990 Apr;6(4):535-42. doi: 10.1089/aid.1990.6.535. PMID 2187503
- [Background] Viscidi R, Ellerbeck E, Garrison L, Midthun K, Clements ML, Clayman B, Fernie B, Smith G. Characterization of serum antibody responses to recombinant HIV-1 gp160 vaccine by enzyme immunoassay. NIAID AIDS Vaccine Clinical Trials Network. AIDS Res Hum Retroviruses. 1990 Nov;6(11):1251-6. doi: 10.1089/aid.1990.6.1251. PMID 1706607
- [Background] Orentas RJ, Hildreth JE, Obah E, Polydefkis M, Smith GE, Clements ML, Siliciano RF. Induction of CD4+ human cytolytic T cells specific for HIV-infected cells by a gp160 subunit vaccine. Science. 1990 Jun 8;248(4960):1234-7. doi: 10.1126/science.2190315.
- [Background] Clerici M, Berzofsky JA, Shearer GM, Tacket CO. Exposure to human immunodeficiency virus (HIV) type I indicated by HIV-specific T helper cell responses before detection of infection by polymerase chain reaction and serum antibodies [corrected]. J Infect Dis. 1991 Jul;164(1):178-82. doi: 10.1093/infdis/164.1.178. PMID 1829105
- [Background] Bollinger RC, Quinn TC, Liu AY, Stanhope PE, Hammond SA, Viveen R, Clements ML, Siliciano RF. Cytokines from vaccine-induced HIV-1 specific cytotoxic T lymphocytes: effects on viral replication. AIDS Res Hum Retroviruses. 1993 Nov;9(11):1067-77. doi: 10.1089/aid.1993.9.1067. PMID 7906131
- [Background] Polydefkis M, Koenig S, Flexner C, Obah E, Gebo K, Chakrabarti S, Earl PL, Moss B, Siliciano RF. Anchor sequence-dependent endogenous processing of human immunodeficiency virus 1 envelope glycoprotein gp160 for CD4+ T cell recognition. J Exp Med. 1990 Mar 1;171(3):875-87. doi: 10.1084/jem.171.3.875. PMID 1968506